CLINICAL TRIAL: NCT06312670
Title: Phase 2 Trial Combining EPI-7386 With Enzalutamide and Androgen Deprivation Therapy for Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: Combining EPI-7386 With Enzalutamide and Androgen Deprivation Therapy for Metastatic Hormone-Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pedro Barata, MD, MSc (Other)
Collaborators: ESSA Pharma Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Barata, MD, MSc, Director, Clinical Genitourinary Medical Oncology Research Program, Prinicipal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2823
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC); Prostate Cancer; Prostate Adenocarcinoma
Keywords: Metastatic Hormone-sensitive Prostate Cancer (mHSPC); Prostate Cancer; Androgen Deprivation Therapy; Prostate adenocarcinoma; Recurrent metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — enzalutamide; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Phase 2, single-arm study composed of 2 stages: in the first stage, 13 subjects diagnosed with mHSPC will be enrolled and treated with EPI-7386 in combination with enzalutamide. If there are 8 or less subjects with a biochemical response at 6 months, then the trial will be suspended. Otherwise, 22 additional subjects will be enrolled and treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPI-7386 + Enzalutamide (Experimental): EPI-7386 at 600 mg twice daily orally with standard of care Enzalutamide at 160 mg, once daily, orally for 36 months of treatment (11 cycles).
  Interventions: Drug: EPI-7386; Drug: Enzalutamide; Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Drug: EPI-7386 — 600 mg orally administered twice daily
Drug: Enzalutamide — 160 mg administered orally once daily, with or without food
Drug: Androgen Deprivation Therapy (ADT) — LHRH agonist/antagonist or orchiectomy

SUMMARY:
The purpose of this study is to study the effects of EPI-7386 in combination with Enzalutamide on participants diagnosed with prostate cancer. The main goals of this study are to evaluate the antitumor activity of EPI-7386 in combination with enzalutamide in metastatic hormone-sensitive prostate cancer (mHSPC), and to evaluate the pharmacokinetics (PK) of EPI-7386 when dosed in combination with enzalutamide. Participants will will take the study drug, EPI-7360, twice a day by mouth and enzalutamide once a day by mouth, alongside clinic visits every two weeks.

DETAILED DESCRIPTION:
EPI-7386 is an investigational drug that works by blocking the androgen receptor at a different site compared to the approved androgen receptor blockers. This may increase the effectiveness of this drug and increase the effectiveness of approved androgen receptor blockers when taken together. EPI-7386 is a new drug; therefore, its effectiveness and safety in prostate cancer patients must be studied before it is approved by the Food and Drug Administration. EPI-7386 is experimental because it is not currently approved by the Food and Drug Administration (FDA). Enzalutamide is approved by the FDA for patients whose prostate cancers has spread after receiving treatment. The hypothesis is that adding EPI-7386 to standard hormone therapy will be more effective in treating cancer compared to usual treatment, with the long term goal of discovering more about hormone therapy as a treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed prostate adenocarcinoma without small cell or neuroendocrine features (please note: >10% small cell or neuroendocrine differentiation will be excluded).
* Subjects must have received no prior second-generation antiandrogen therapies for this disease. Androgen deprivation with LHRH agonist/antagonist therapy or history of bilateral orchiectomy that started less than 12 weeks before study enrollment is allowed.
* Subjects may have either de novo or recurrent metastatic disease. Presence of metastatic disease at study entry documented by 1 or more lesions - bone, lymph node, soft tissue, or visceral metastases - observed by any imaging technique.
* Age >18 years. This study will be limited to adults only.
* Evidence of metastatic disease by conventional CT of chest, abdomen, and pelvis, and bone scans, OR Positron emission tomography (PET) scan, OR MRI.
* ECOG performance status of 0 to 2.
* Subjects must have normal organ and marrow function as defined below:

  * Absolute neutrophil count >1000/μL; platelet count >100 000/μL; hemoglobin >8.5 g/dL) at screening. Note: Subjects must not have received any growth factors within 7 days or blood transfusions within 14 days prior to the hematologic laboratory values obtained at screening).
  * Total bilirubin (TBIL) <2 × the upper limit of normal (ULN) at screening, except subjects with documented Gilbert syndrome who must have a TBIL <3 mg/dL
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <5 × ULN at screening
  * Creatinine clearance ≥45 mL/min and/or estimated glomerular filtration rate (eGFR) ≥30
  * Albumin >30 g/L (3.0 g/dL) at screening
* Subjects receiving bisphosphonates or other approved bone-targeting therapy (e.g., denosumab) must be on a stable dose for at least 28 days before the start of study treatment.
* Radiation therapy is allowed at any time, as deemed appropriate by the treating investigator.
* Subjects of child-producing potential agree to use highly effective contraceptive methods (i.e., barrier contraception measures such as a male condom with spermicide during intercourse) and avoid sperm donation during the study treatment and for 3 months after the last dose of study treatment. A man is considered to be of child-producing potential, unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy. Partners of participants must also practice approved forms of birth control.
* Subjects must have the ability to understand and the willingness to sign a written informed consent form (ICF).
* Members of all races and ethnic groups are eligible for this trial. At least ≥ 20% of enrolled subjects must be of African American descent. (self-reported).

Exclusion Criteria:

* Evidence of mCRPC.
* Receipt of any other investigational agents.
* Diagnosis of another clinically significant malignancy within the previous 3 years other than curatively treated non-melanomatous skin cancer or superficial urothelial carcinoma and other in situ or noninvasive malignancies, as determined by the PI or CoPI.
* Gastrointestinal issues affecting absorption (e.g., gastrectomy).
* Known history of seizure or conditions that may predispose the subject to seizure, including brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain metastases, or brain arteriovenous malformation. Subjects with brain metastases/central nervous system (CNS) disease that are treated prior to enrollment will be allowed in this clinical trial.
* Known or suspected hypersensitivity to any components of the formulation used for EPI-7386 or enzalutamide.
* Use of compounds known to be strong inducers of CYP3A within 30 days prior to start of study drug treatment, and strong inhibitors of CYP2C8 within 14 days of the first dose of study treatment.
* Use of narrow therapeutic index sensitive CYP2C8 substrates (e.g., daprobustat, dasabuvir, repaglinide, paclitaxel) or sensitive substrates for CYP3A.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations considered by the Investigator to limit compliance with study requirements.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Biochemical response rate | Post-intervention at Week 4
  Defined as prostate-specific antigen (PSA) undetectable (<0.2 ng/mL) at 6 months after treatment. The true BRR for the study population will be estimated based on the number of biochemical responses using a binomial distribution, and its confidence interval (CI) will be estimated using Wilson's method.
PSA progesterone-free survival (PFS) | Post-intervention at Week 4
  Progression free survival (PFS) is measured from the date of the start of the treatment to the date of progression or death and is censored at the date of last followed for those that have not progressed
Radiographic PFS (rPFS) | Post-intervention at Week 4
  Progression free survival (PFS) is measured from the date of the start of the treatment to the date of progression or death and is censored at the date of last followed for those that have not progressed
ORR (confirmed) | Post-intervention at Week 4
  Objective response rate (ORR)

SECONDARY OUTCOMES:
AUC0-24 | Beginning of treatment day 1, at week 2, week 4, week 6
  Plasma area under the concentration-time curve from time zero to 24 hours (AUC0-24)
Maximum concentration (Cmax) | Beginning of treatment day 1, at week 2, week 4, week 6
  Total Maximum concentration
Predose Plasma Concentration | Beginning of treatment day 1, at week 2, week 4, week 6
  Observed predose plasma concentration during multiple dosing (Ctrough)
Time to reach Cmax (Tmax) | Beginning of treatment day 1, at week 2, week 4, week 6
  Time it takes to reach maximum concentration
Terminal elimination half-life | Beginning of treatment day 1, at week 2, week 4, week 6
  Apparent terminal elimination half-life (t½), whenever feasible to calculate
Volume of distribution at steady state after extravascular administration | Beginning of treatment day 1, at week 2, week 4, week 6
  Apparent volume of distribution at steady state after extravascular administration (Vss/F)
Clearance after extravascular administration | Beginning of treatment day 1, at week 2, week 4, week 6
  Apparent clearance after extravascular administration.
Treatment-emergent adverse events | Post-intervention at Week 4
  Treatment-emergent adverse events (TEAEs) (characterized by type, frequency, severity, timing, seriousness, and relationship to study treatment)
Rate of abnormalities in clinical laboratory parameters | Baseline, 2 weeks, 11 weeks, and 20 weeks after beginning treatment
  The presenece of abnormalities in clinical laboratory parameters will be measured and characterized by type, frequency, severity, timing, seriousness, and relationship to study treatment.
Rate of abnormalities in vital sign measurements | Post-intervention at Week 4
  The presence of abnormalities in vital sign measurements will be measured and characterized by type, frequency, severity, timing, seriousness, and relationship to the study treatment.
Rate of abnormalities in electrocardiograms (ECGs) | At screening and beginning of treatment on day 1 of cycle 1 (each cycle is 14 days)
  The presence of abnormalities in ECGs will be measured and characterized by type, frequency, severity, timing, seriousness, and relationship to the study treatment.
Changes in Eastern Cooperative Oncology Group (ECOG) performance status | Post-intervention at Week 4
  Changes in ECOG performance status. The ECOG performance status relies on a scale with scores ranging from 0-5, where 0 indicates the highest function, and 5 indicates lowest function.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Barata, MD, MSc, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Christopher Wee, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed from the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Compiled and analyzed participant data will be published upon study completion.
Access Criteria: Link to be provided at time of article publication.

REFERENCES:
- [Derived] Jang A, Fowler P, Helminiak K, Kumar HLS, Pasucal J, Delong V, Zhong JY, Jindal T, Grier AL, Patel RR, Hislop M, Cesano A, Villaluna K, Younginger B, Wolff K, Richey K, Bray J, Garcia H, Adamowicz T, Reese A, Nizam A, Gupta S, Wee CE, Margevicius S, Fu P, Mendiratta P, Sheng IY, Brown JR, Garcia JA, Barata PC. EXTRA-PC: A phase II trial of masofaniten (EPI-7386) and enzalutamide for patients with treatment-naive metastatic hormone-sensitive prostate cancer. Oncologist. 2025 Dec 30:oyaf434. doi: 10.1093/oncolo/oyaf434. Online ahead of print. PMID 41467749